CLINICAL TRIAL: NCT04797663
Title: Clinical and Dermoscopic Evaluation of Long-pulsed 1064 nm Nd-YAG Laser Versus Trichloroacetic Acid 20% in Treatment of Keratosis Pilaris
Brief Title: Long-pulsed 1064 nm Nd-YAG Laser Versus TCA 20% in Treatment of Keratosis Pilaris
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Saadi, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: las177
Record Dates: First submitted 2021-03-06; First posted 2021-03-15 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Keratosis Pilaris
MeSH Terms: conditions — Burnett Schwartz Berberian syndrome | interventions — Lasers, Solid-State; Lasers; Trichloroacetic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Nd-YAG laser (Active Comparator): laser hair removal
  Interventions: Device: Nd-YAG laser
- TCA 20% (Experimental): chemical peel
  Interventions: Drug: TCA 20%

INTERVENTIONS:
Device: Nd-YAG laser — laser hair removal device
  Other Names: 1064 nm laser
  Arms: Nd-YAG laser
Drug: TCA 20% — chemical peel
  Other Names: Trichloroacetic acid
  Arms: TCA 20%

SUMMARY:
Keratosis pilaris (KP) is a common disorder of keratinization. There are different treatment modalities for KP with variable results. Nd:YAG laser and chemical peels are among these treatment modalities, however, there is no enough evidence in the literature regarding their efficacy. The aim of this study is to assess and compare the efficacy of long pulsed Nd:YAG laser and trichloreacetic acid 20% in treatment of keratosis pilaris.

DETAILED DESCRIPTION:
Keratosis pilaris (KP) is a genetic disorder of keratinization of hair follicles of skin. It's a very common benign condition that manifests as small, rough folliculocentric keratotic papules, often described as chicken bumps, chicken skin or goose-bumps, in characteristic areas of body, particularly the outer upper arms and thighs.

Trichloreacetic acid (TCA) is a type of chemical peels that is derived from acetic acid by the chlorination of 3 hydrogen ions. It can induce coagulative necrosis of proteins and cells. The depth of action depends on various factors e.g the number of layers applied and its combination with substances that potentiate its action.

Nd: YAG laser is a type of hair removing devices that operates at wave length of 1064nm. This wave length allows for less absorption at the epidermis. It is less absorbed by melanin, which leads to lower side effect and better tolerance but less efficacy in dark skinned patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years with KP.
* Patients with KP affecting back of the trunk, arms, thighs, forearms, legs and buttocks.

Exclusion Criteria:

* Pregnant or lactating females.
* Patients who had performed any laser treatment for KP within 6 months prior to the study.
* Patients with history of oral retinoids within 3 months prior to the study.
* Patients with history of hypertrophic scars or keloids.
* Patients who used any topical treatment one month prior to the session.
* Patients with acne affecting the same sites of keratosis pilaris.
* Patients with active skin diseases affecting the area involved with KP e.g. folliculitis and eczema.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2021-07-18 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Change of clinical and dermoscopic scores of KP with Nd-YAG laser | 4 months
  the change in roughness and color of KP by clinical score after 4 sessions of Nd-YAG laser. the score ranges from 0-4. where 0 is no change and 4 is excellent improvement
Change of clinical and dermoscopic scores of KP with TCA 20% | 4 months
  the change in roughness and color of KP by clinical score after 4 sessions of TCA 20% peel. the score ranges from 0-4. where 0 is no change and 4 is excellent improvement

SECONDARY OUTCOMES:
safety and tolerability of Nd-YAG laser and TCA 20% in treatment of KP: adverse events | 4 months
  adverse effects of treatment modalities, if any

CONTACTS AND LOCATIONS:
Overall Officials: Akmal Saad, professor, Principal Investigator — Cairo University
Locations (1):
- Kasr Alainy, Cairo, Egypt

REFERENCES:
- [Derived] Hassan AS, Abdel Aziz M, Saadi DG. Clinical and Dermoscopic Evaluation of Trichloroacetic Acid 20% Versus Long-Pulsed 1064-nm Nd-YAG Laser in the Treatment of Keratosis Pilaris. Dermatol Surg. 2022 Aug 1;48(8):838-842. doi: 10.1097/DSS.0000000000003488. Epub 2022 Jun 15. PMID 35917264